## **INFORMED CONSENT**

## Using Retrospective and Real-Time Physical Activity Tracking to Predict Risk of Sunburn in Outdoor Exercisers on Strava

NCT04977700

06/22/2020

## Research Subject Information Sheet Collection of Retrospective Activity Data

TITLE: Using Retrospective and Real-Time Physical Activity Tracking to

Predict Risk of Sunburn in Outdoor Exercisers on Strava

**PROTOCOL NO.:** 1R21CA241637-01A1

WIRB® Protocol #20201655

**SPONSOR:** National Cancer Institute (NCI)

**INVESTIGATOR:** David Buller, PhD

1667 Cole Blvd, Ste 225 Golden, Colorado 80401

STUDY-RELATED

PHONE NUMBER(S): David Buller, PhD

303-565-4321

You are being asked to be in a research study. The study's goal is to develop, produce, and test a smartphone application to develop new mHealth strategies to reduce the epidemic of skin cancer in the United States. In addition, the *Strava Sun (SS)* app will provide physically active Americans a healthy lifestyle behavior and real-time advice on sun safety, when and where they need it.

Your participation will NOT involve answering survey questions or actively participating in the program. If you agree to participate you will provide authentication to collect one year of your retrospective activity data through *Strava*. We will not collect your current activity data. The data being collected and what it will be used for will be detailed in the authentication. Your participation will end at the end of one year.

Eligibility requirements include: 1) having at least 156 activities uploaded in one year of *Strava* use; 2) providing authentication. You will be entered to win one of ten \$50 gift cards for allowing access to your data.

There is a slight risk that your confidentiality may be compromised.

You will be told about any new information that might change your decision to be in this study.

You may not receive a direct benefit if you agree to participate. However, people in the future may benefit from the information obtained from this research.

This is not a treatment study and your alternative is to not participate in this study.

Contact David Buller, PhD at 303-565-4321 for questions, concerns or complaints about the research or if you think you have been harmed as a result of joining this research. Contact the Western Institutional Review Board (WIRB) if you have questions about your rights as a research subject, concerns, complaints or input: 1-800-562-4789. WIRB is a group of people who perform independent review of research.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

The study staff may share the records generated from this research with the sponsor, regulatory agencies such as Department of Health and Human Services (DHHS) or the US Food and Drug Administration (FDA) and the IRB. This information is shared so the research can be conducted and properly monitored. The people receiving this information may not be required to protect it and your information may be redisclosed without your permission. If you do not provide permission to use your information you cannot be in the study.

There is a possibility that identifiers might be removed from the identifiable private information, and after such removal, the information may be used for future research studies or distributed to another investigator for future research studies without additional informed consent from the subject or the legally authorized representative.

This permission will not end unless you cancel it. You may cancel it by sending written notice to the Principal Investigator at <u>303-565-4321</u> or dbuller@kleinbuendel.com. Any information collected before you withdraw may still be used.

Your decision to be in this study is voluntary. You will not be penalized or lose benefits to which you are otherwise entitled if you decide not to participate or if you decide to stop participating.

Your part in this study may be stopped at any time by the study doctor or the sponsor without your consent for any reason, including:

- if it is in your best interest;
- you do not consent to changes made in the study plan;
- or for any other reason.

| _ I agree to participate in this study |
|---------------------------------------------|
| I do not agree to participate in this study |